CLINICAL TRIAL: NCT00734123
Title: Early Detection of Atherosclerosis in the Primary Care Setting: a Randomized Trial to Assess the Efficacy of a Novel Strategy in the Primary Prevention of Cardiovascular Diseases.
Brief Title: Early Detection of Atherosclerosis: a Randomized Trial in the Primary Prevention of Cardiovascular Diseases.
Acronym: PRIMARIA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Arnau de Vilanova (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Elvira Fernandez, Hospital Arnau de Vilanova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UDETMA_08; UDETMA_2008_001
Record Dates: First submitted 2008-08-11; First posted 2008-08-14 (Estimated); Last update posted 2008-08-14 (Estimated); Status verified 2008-08

CONDITIONS: Atherosclerosis; Cardiovascular Diseases
Keywords: Atherosclerosis; Cardiovascular Prevention; Carotid Intima-Media Thickness; Ankle-Brachial Index
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases | interventions — Simvastatin; Atorvastatin; Enalapril; Angiotensin-Converting Enzyme Inhibitors; Diuretics; Aspirin; Clopidogrel; Rimonabant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants assigned to the intensive arm (1) will be targeted to specified therapeutic aims (concerning lipids, blood pressure and antiplatelets)according to the results of carotid ultrasound and ankle-brachial index.
  Interventions: Drug: Simvastatin or Atorvastatin; Drug: Enalapril; Drug: Aspirin or clopidogrel; Drug: Rimonabant
- 2 (Active Comparator): Participants assigned to control group (2) will be followed according to the clinical standard of care.
  Interventions: Drug: Rimonabant

INTERVENTIONS:
Drug: Simvastatin or Atorvastatin — Simvastatin 10-40 mg or Atorvastatin 20-40 mg will be prescribed according to LDL cholesterol reduction target.
  Other Names: Simvastatin 10-40.; Atorvastatin 20-40.
  Arms: 1
Drug: Enalapril — Enalapril 10 mg/day will be prescribed as the initial treatment. Doses and adding drugs will be titrated accordingly
  Other Names: ACE inhibitors.; ACE + diuretic
  Arms: 1
Drug: Aspirin or clopidogrel — Aspirin 100 mg or clopidogrel 75 mg/ per day
  Other Names: Antiplatelets
  Arms: 1
Drug: Rimonabant — In both arms, we will follow the standard clinical care in terms of treatments, as far as obesity and diabetes mellitus is concerned.
  Drugs will be prescribed as the standard clinical care
  Other Names: Rimonabant is allowed.

SUMMARY:
The incidence of cardiovascular diseases is still high and further efforts should be done in primary prevention. The main objective is to quantify the burden of subclinical atherosclerosis using non-invasive techniques,and to study the impact of this assessment and consequent treatment in the progression of atherosclerosis and in the incidence of cardiovascular diseases.

DETAILED DESCRIPTION:
We will perform non-invasive techniques (carotid Intima-Media Thickness, CAC score and ankle-brachial index) to individuals at intermediate cardiovascular risk.With these results, we will classify participants in: no atherosclerosis, mild, moderate and severe atherosclerosis, and therapeutic targets will be set according to pre-defined algorithms. The end-point will be the course of atherosclerosis measured by cIMT/CAC score (2 years) and the incidence of CVD at 5 years of follow-up.

ELIGIBILITY:
Inclusion Criteria

One or more of the following:

* Familiar History of early-onset cardiovascular disease (male < 55 or female < 65).
* Type 2 Diabetes mellitus or type 1 with microalbuminuria.
* Essential High Blood Pressure.
* Chronic Kidney Disease.
* Primary hyperlipidemia.

The presence of two or more of the following:

* Current smoker.
* Physical inactivity.
* High blood pressure (recently diagnosed).
* Abdominal perimeter: > 102 cm. males; > 88 cm. females.
* Total cholesterol > 240 mg/dL.
* HDL cholesterol ≤ 40 mg/dL males, ≤ 50 mg/dL females.

Exclusion Criteria:

* Age < 40 or > 74 years old.
* Previous Cardiovascular Event.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2948 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-04 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Carotid Intima-Media Thickness progression/regression | 2 years

SECONDARY OUTCOMES:
Cardio and cerebrovascular eventS | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Elvira Fernandez, MD,PhD, Principal Investigator — Hospital Arnau de Vilanova
Locations (1):
- Hospital Arnau de Vilanova, Lleida, Catalonia, Spain